CLINICAL TRIAL: NCT01472796
Title: Vitamin D Augmentation of Tekturna (Aliskiren) in Hypertension (VDATH)
Brief Title: Vitamin D Augmentation of Tekturna (Aliskiren) in Hypertension
Acronym: VDATH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, John M. Flack, Chairman, Dept. of Internal Medicine, Wayne State University, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100AUS41T
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: African American; Vitamin D deficient
MeSH Terms: conditions — Hypertension | interventions — Cholecalciferol; aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tekturna (Aliskirin) with vit. D supplementation (Active Comparator): Tekturna (Aliskiren) 300mg daily and vitamin D supplementation (50,000 IU)every other week.
  Interventions: Dietary Supplement: Vitamin D (cholecalciferol)
- Tekturna (Aliskiren) with placebo (Placebo Comparator): Tekturna (Aliskiren) 300mg per day supplemented with placebo (vitamin D)
  Interventions: Drug: Tekturna(Aliskiren) plus placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D (cholecalciferol) — Tekturna (Aliskirin) 300 mg per day supplemented with 50,000 IU Vitamin D every other week x 8 weeks
  Other Names: Tekturna (Aliskirin); cholecalciferol
  Arms: Tekturna (Aliskirin) with vit. D supplementation
Drug: Tekturna(Aliskiren) plus placebo — Aliskiren 300 mg per day supplemented with placebo
  Other Names: Tekturna (Aliskirin)
  Arms: Tekturna (Aliskiren) with placebo

SUMMARY:
In this research study, the goal is to find out if a currently FDA-approved medication called Tekturna(Aliskiren) along with the addition of Vitamin D will lower blood pressure and improve heart function in the African American population. High blood pressure occurs earlier in life in African Americans, is more severe, and is associated with greater organ damage in relation to uncontrolled hypertension. Having low levels of Vitamin D is also very common in the African American population. Research has shown that there may be a link between low Vitamin D levels and the ability of high blood pressure medications to be fully effective.

DETAILED DESCRIPTION:
The overarching hypothesis is that African Americans with hypertension have an overactive RAS (Renin Angiotensin System) in the body that is responsible for internally regulating blood pressure. Many blood pressure medications change regulation of the RAS system in order to keep blood pressure down. The purpose of this research study is to determine whether or not African American adults with hypertension have an overactive RAS system due to Vitamin D deficiency, resulting in the inability of the medication Tekturna to lower blood pressure. In this study, all participants will receive 300mg of Tekturna per day. Additionally half of the participants will randomly be selected to receive either 50,000 IU of Vitamin D (in its cholecalciferol form) orally once every other week or a vitamin D placebo once every other week. There will be 4 study visits over 18 weeks and follow up phone calls every two weeks for the duration of the study.

Specific Aims:

To demonstrate in African American Hypertensives consuming a calcium replete diet that Tekturna + Vitamin D will lower blood pressure more than Tekturna + placebo.

To demonstrate in African American hypertensives consuming a calcium replete diet that albuminuria will be lowered more with Tekturna + Vitamin D versus Tekturna + placebo.

To demonstrate in African American hypertensives consuming a calcium replete diet that Tekturna + Vitamin D will improve measures on non-invasively measured vascular function (peripheral vascular resistance, augmentation index, carotid-femoral pulse wave velocity and central aortic pressure) more than Tekturna + placebo.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30-74
* Systolic Blood Pressure 140-159 mm Hg and Diastolic Blood Pressure <100 OR Diastolic Blood Pressure 90-99mm Hg and Systolic Blood Pressure <160mm Hg
* Vitamin D deficiency: Serum 25-OH D >= 10 ng/ml (25 nmol/L) to < 20 ng/ml (50 nmol/L)
* Not using any antihypertensive medication(s) for the previous 3 months

Exclusion Criteria:

* Cancer(other than skin) known HIV or other medical condition that might limit life expectancy.
* Pregnant or nursing
* Know adverse reactions to DRI's
* Hepatitis or liver enzyme elevations > 1.5x normal
* Estimated glomerular filtration rate (EGFR) <50 ml/min/1.7m2
* Diabetes Mellitus
* Serum calcium > 10.5 mg/dl or history of hypercalcemia
* History of primary hyperparathyroidism
* Sarcoidosis or other granulomatous disease
* Taking > 500 mg/d of supplemental elemental calcium
* Taking any drugs that decrease absorption of vitamin D, ex:xenical
* Taking the drug cyclosporine
* Taking any antihypertensive medications in the previous 3 months
* History of kidney stones
* Planning to move > 50 miles in the next 9 months

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change in Ambulatory Systolic Blood Pressure | from baseline (Week 10) to Week 18

SECONDARY OUTCOMES:
Change in ambulatory diastolic blood pressure | from baseline (Week 10) to Week 18
Change in cuff systolic blood pressure | from baseline (Week 10) to Week 18
Change in cuff diastolic blood pressure | from baseline (week 10) to Week 18
Change in Urinary albumin:creatinine ratio | from baseline (week 10) to Week 18
Change in plasma isoprostanes | from baseline (week 10) to Week 18
Change in urinary nitric oxide metabolites | from baseline (week 10) to Week 18
Change in plasma renin activity | from baseline (week 10) to Week 18
Change in urinary angiotensinogen | from baseline (week 10) to Week 18
Change in non-invasively obtained measures of vascular function | from baseline (week 10) to Week 18

CONTACTS AND LOCATIONS:
Overall Officials: John M Flack, M.D., M.P.H., Principal Investigator — Wayne State University, TRaCE Research Group
Locations (1):
- Wayne State University, 4201 St. Antoine, Detroit, Michigan, United States